CLINICAL TRIAL: NCT06575439
Title: An Observational Study of Predictors and Outcomes of Lung Cancer in Never-smokers in the UK
Acronym: OLIVE
Status: Recruiting | Type: Observational
Sponsor: University College London Hospitals (Other)
Responsible Party: Principal Investigator, Neal Navani, Professor of Respiratory Medicine, University College, London
Other Study IDs: 159292
Record Dates: First submitted 2024-08-21; First posted 2024-08-28 (Actual); Last update posted 2024-12-12 (Actual); Status verified 2024-12

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The goal of this observational study is to improve the early detection of lung cancer in adults who have smoked less than 100 tobacco cigarettes ("never-smokers") in the United Kingdom. The main questions it aims to answer are:

* To describe characteristics such as demographics, co-morbidities and environmental exposures
* To describe participant pathways including presentation mode and symptoms to understand if earlier diagnosis would be possible
* To describe participant outcomes such as cancer stage, treatment and mortality
* To quantitatively or qualitatively measure modifiable and non-modifiable factors that may be associated with LCINS including environmental measures, blood tests and genomic data.

Participants will currently have no change to their usual care.

ELIGIBILITY:
Inclusion Criteria:

* All adult participants from age of 18 who are diagnosed or treated with primary lung cancer through radiology or histology at any participating study site

Exclusion Criteria:

* Participants who have ever smoked cigarettes or tobacco will be excluded; this is defined as:

  * More than 100 cigarettes or 75g tobacco in their lifetime
  * Those who have received a prescription for nicotine replacement therapy
* For prospective participants, those who cannot consent will be excluded

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will aim to recruit participants who have been diagnosed or treated with primary lung cancer at any participating study site.
Sampling Method: Non-Probability Sample
Enrollment: 225 (Estimated)
Dates: Start 2024-09-17 (Actual); Primary Completion 2029-09 (Estimated); Study Completion 2029-09 (Estimated)

PRIMARY OUTCOMES:
Demographics, comorbidities and environmental exposures of participants | Comorbidities and environmental exposures at diagnosis (approximately up to 156 weeks prior to diagnosis)
  From review of electronic health records
Participant pathways including presentation mode and symptoms | Presentation mode and symptoms at time of diagnosis (approximately up to 52 weeks prior to diagnosis)
  From review of electronic health records

SECONDARY OUTCOMES:
Participant outcomes such as cancer stage, treatment, mortality | Cancer stage at time of diagnosis, treatment and mortality through study completion (likely 5 years)
  From review of electronic health records
Measurement of modifiable and non-modifiable factors associated with LCINS | Through study completion (likely 5 years)
  To be determined

CONTACTS AND LOCATIONS:
Locations (1):
- University College London Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No
No individual participant data will be made available to non-study researchers (as per current ethics approval).